CLINICAL TRIAL: NCT01203787
Title: Multicenter, Randomized Pilot Study of the Effect of Sorafenib Dosing Schedule on Tolerability and Drug Delivery
Brief Title: Sorafenib Dose Ramp-Up in Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2010-19
Record Dates: First submitted 2010-09-10; First posted 2010-09-16 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; HCC; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sorafenib Standard Dosing Regimen (Active Comparator): Sorafenib 400 mg (2 tablets of 200 mg) twice daily until end of treatment or week 24
  Interventions: Drug: Sorafenib Ramp-Up Regimen
- Sorafenib Ramp-Up Regimen (Experimental): 200 mg daily from Day 0-Day 13 200 mg twice daily from Day 14-Day 20 600 mg daily from Day 21-Day 27 400 mg twice daily beginning Day 28 until end of treatment or Week 24
  Interventions: Drug: Sorafenib Standard Dosing Regimen

INTERVENTIONS:
Drug: Sorafenib Standard Dosing Regimen — Sorafenib 400 mg twice daily until wk 24 or end of treatment
  Other Names: Nexavar(Bay43-9006)
  Arms: Sorafenib Ramp-Up Regimen
Drug: Sorafenib Ramp-Up Regimen — 200 mg daily, Day 0-Day 13 200 mg twice daily, Day 14-Day 20 600 mg daily, Day 21-Day 27 400 mg twice daily, Day 28 until end of treatment400 mg twice daily
  Other Names: Nexavar (Bay43-9006)
  Arms: Sorafenib Standard Dosing Regimen

SUMMARY:
Open-label study to evaluate the safety and tolerability of Sorafenib dose ramp-up (starting at a lower dose and then gradually increasing the dose) versus standard Sorafenib dosing in subjects with unresectable and/or metastatic hepatocellular carcinoma.

DETAILED DESCRIPTION:
This is an open-label study that investigates the impact of a dose ramp-up strategy for sorafenib in patients with HCC. Clinical trial and post-marketing data suggest that sorafenib dose reductions and discontinuations due to adverse events are common and limit the drug's effectiveness. It is our hypothesis that a dose escalation strategy for sorafenib will improve the tolerability and allow a greater percentage of patients to remain on drug. The primary end-point of the study is the total accumulated and median daily dose of sorafenib delivered at month 2 and 4.

ELIGIBILITY:
Inclusion Criteria:

* HCC must be unresectable and/or metastatic
* CPT score <9 at the time of screening (that is all Child A and Child B with a score of 7 or 8)
* Age 20-75 years
* Signed informed consent
* EGD for variceal screening performed as per standard of care prophylaxis with non-selective beta-blockers or ligation
* ECOG Performance Status ≤ 2.
* Adequate bone marrow, liver and renal function as assessed by the following:

  1. Hemoglobin > 8.5 g/dl
  2. Absolute neutrophil count (ANC) > 1,500/mm3
  3. Platelet count > 50,000/mm3
  4. Total bilirubin < 3 mg/dl
  5. ALT and AST ( < 5 x ULN)
  6. Creatinine < 1.5 times ULN
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and non-surgically sterile men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* INR< 2.3. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Life expectancy of at least 24 weeks

Exclusion Criteria:

* Absence of informed consent
* Child-Pugh score >9
* ECOG PS >2
* Active alcohol dependence per PI discretion
* History of organ or bone marrow transplant
* Plans to relocate from the study center within the period of the trial
* Pregnancy or breastfeeding
* Contraindications to sorafenib

  1. Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
  2. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
  3. Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
  4. Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection
* Active clinically serious infection > CTCAE Grade 2.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Bleeding

  1. Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
  2. Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
  3. Evidence or history of bleeding diathesis or coagulopathy
* Serious non-healing wound, ulcer, or bone fracture.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks prior to first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-12; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Nelson, MD, Principal Investigator — University of Florida
Locations (9):
- United States (9):
  - University of Florida Hepatology, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Florida Hospital Transplant Center, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Texas Health Science Center Houston, Houston, Texas
  - Brooke Army Medical Center, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sorafenib Standard Dosing Regimen | Sorafenib Ramp-Up Regimen
Started | 63 | 57
Completed | 32 | 30
Not Completed | 31 | 27
Not completed — Death | 12 | 10
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Sorafenib Ramp-Up Regimen: 200 mg daily from Day 0-Day 13, 200 mg twice daily from Day 14-Day 20, 600 mg daily from Day 21-Day 27, 400 mg twice daily beginning Day 28 until end of treatment or Week 24
- Total: Total of all reporting groups
Arm/Group | Sorafenib Standard Dosing Regimen | Sorafenib Ramp-Up Regimen | Total
Number analyzed (Participants) | 63 | 57 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 00 | 00 | 0
  Between 18 and 65 years | 39 | 30 | 69
  >=65 years | 24 | 27 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (6.8) | 63.5 (7.5) | 62.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 51 | 47 | 98
Region of Enrollment [Number; unit: participants]
  United States | 63 | 57 | 120

OUTCOME MEASURES:

1. Primary Outcome: Total (Cumulative) Dose Delivery of Sorafenib
Description: This outcome measure table shows the median cumulative dose delivered to the subjects randomized to the standard dosing regimen (N=63) and ramp-up regimen (N=57) at 4 months of treatment.
Time Frame: 4 months-1/12/2010-1/27/14
Measure: Median (Full Range); unit: mg
Arm/Group | Sorafenib Standard Dosing Regimen | Sorafenib Ramp-Up Regimen
Number analyzed (Participants) | 63 | 57
mg | 49800 [800 to 107600] | 38000 [800 to 92400]
Statistical Analysis 1: Comparison: Sorafenib Standard Dosing Regimen vs Sorafenib Ramp-Up Regimen; Test type: Superiority or Other; p = 0.0262, Wilcoxon rank sum test

2. Secondary Outcome: Safety and Efficacy of Sorafenib Dosing Regimens
Description: Safety of Sorafenib was assessed by the frequency and severity of adverse events according to NCI-CTCAE grading
Time Frame: Baseline-End of Treatment (11/22/2010-3/10/2014)
Population: The total number of CTCAE (Common Terminology Criteria) grade 3 adverse events was collected for each dosing regimen
Measure: Number; unit: Grade 3 adverse events
Arm/Group | Sorafenib Standard Dosing Regimen | Sorafenib Ramp-Up Regimen
Number analyzed (Participants) | 63 | 57
Grade 3 adverse events | 92 | 101

3. Secondary Outcome: Safety of Dosing Regimens as Assessed by the Frequency and Severity of Adverse Events According to National Cancer Institute- CTCAE
Description: The total number of CTCAE (Common Terminology Criteria) grade 4 adverse events was collected for each dosing regimen beginning at baseline until Week 24/Early Termination Visit.
Time Frame: 11/22/2010-3/10/2014
Measure: Number; unit: Grade 4 adverse events
Arm/Group | Sorafenib Standard Dosing Regimen | Sorafenib Ramp-Up Regimen
Number analyzed (Participants) | 63 | 57
Grade 4 adverse events | 19 | 15

4. Secondary Outcome: Frequency and Severity of Adverse Events According to National Cancer Institute- CTCAE
Description: The total number of CTCAE (Common Terminology Criteria) grade 5 adverse events was collected for each dosing regimen beginning at baseline through 6 months of treatment.
Time Frame: 11/22/2010-3/10/2014
Measure: Number; unit: Grade 5 Adverse Events
Arm/Group | Sorafenib Standard Dosing Regimen | Sorafenib Ramp-Up Regimen
Number analyzed (Participants) | 63 | 57
Grade 5 Adverse Events | 9 | 8

5. Primary Outcome: Cumulative Dose of Sorafenib
Description: Table below shows mean cumulative dose of sorafenib for each of the dosing regimens.
Time Frame: 11/22/2010-1/27/14
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Sorafenib Standard Dosing Regimen | Sorafenib Ramp-Up Regimen
Number analyzed (Participants) | 63 | 57
mg | 53692 (33411) | 41523 (28783)

6. Secondary Outcome: Number of Subjects With Dose Interruptions
Time Frame: Baseline-End of Treatment (11/22/2010-3/10/2014)
Measure: Number; unit: participants
Arm/Group | Sorafenib Standard Dosing Regimen | Sorafenib Ramp-Up Regimen
Number analyzed (Participants) | 63 | 57
participants | 29 | 20

7. Secondary Outcome: Number of Subjects With Dose Reductions
Time Frame: 11/22/2010-3/10/2014
Measure: Number; unit: participants
Arm/Group | Sorafenib Standard Dosing Regimen | Sorafenib Ramp-Up Regimen
Number analyzed (Participants) | 63 | 57
participants | 40 | 34

ADVERSE EVENTS:
Time Frame: Adverse events were collected during 6 months of treatment. First subject randomized 8/29/2011 and last subject completed 6 months of treatment on 3/10/14.
Arm/Group | Sorafenib Standard Dosing Regimen | Sorafenib Ramp-Up Regimen
Serious Adverse Events (participants affected / at risk) | 16/63 | 13/57
Other Adverse Events (participants affected / at risk) | 62/63 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Standard Dosing Regimen (N=63) | Sorafenib Ramp-Up Regimen (N=57)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Acute congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Ascites (Hepatobiliary disorders) | 1 (1) | 1 (2)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Blurred vision (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Decompensated liver failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Deterioration of condition (General disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Encephalopathy (Hepatobiliary disorders) | 6 (6) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 3 (3) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Liver failure (Hepatobiliary disorders) | 0 (0) | 4 (4)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Post-embolization syndrome (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Spontaneous bacterial perotinitis (Infections and infestations) | 1 (1) | 0 (0)
Syncopal episode (General disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Unsteady gait (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Upper gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Standard Dosing Regimen (N=63) | Sorafenib Ramp-Up Regimen (N=57)
abdominal bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal cramps (Gastrointestinal disorders) | 0 (0) | 5 (6)
abdominal pain (Gastrointestinal disorders) | 17 (22) | 21 (26)
abscess (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
allergic rhinitis (Immune system disorders) | 1 (1) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 13 (13) | 7 (7)
ammonia elevation (Hepatobiliary disorders) | 2 (2) | 0 (0)
amylase elevation (Gastrointestinal disorders) | 7 (11) | 6 (6)
anemia (Blood and lymphatic system disorders) | 18 (26) | 16 (19)
ankle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
anorexia (Gastrointestinal disorders) | 17 (20) | 13 (13)
anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
aortic stenosis (Cardiac disorders) | 1 (1) | 0 (0)
arm paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
arthralgias (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (4)
ascites (Hepatobiliary disorders) | 9 (9) | 9 (10)
asterexis (Hepatobiliary disorders) | 0 (0) | 1 (1)
ast elevation (Hepatobiliary disorders) | 1 (1) | 0 (0)
atypical chest pain (Cardiac disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
bacteuria (Renal and urinary disorders) | 0 (0) | 1 (1)
bezoar (Gastrointestinal disorders) | 1 (1) | 0 (0)
bleeding gums (General disorders) | 4 (5) | 0 (0)
blister (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
blurred vision (Eye disorders) | 0 (0) | 3 (3)
bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1)
chest pain (Cardiac disorders) | 0 (0) | 4 (4)
chills (General disorders) | 1 (1) | 2 (2)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
cholelithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
cold intolerance (Endocrine disorders) | 1 (1) | 0 (0)
collar bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
conjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0)
conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 4 (4) | 6 (7)
contusion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
creatinine elevation (Renal and urinary disorders) | 1 (1) | 0 (0)
decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dehydration (General disorders) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 6 (6) | 1 (1)
Diabetic neuropathy (Endocrine disorders) | 1 (1) | 0 (0)
diabetes (Endocrine disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 24 (30) | 23 (28)
diminished breath sounds (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
direct hyperbilirubinemia (Blood and lymphatic system disorders) | 24 (44) | 30 (51)
dizziness (Nervous system disorders) | 2 (2) | 2 (2)
dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
dysgeusia (Gastrointestinal disorders) | 0 (0) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
dysphagia (Gastrointestinal disorders) | 1 (2) | 1 (1)
dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 8 (8)
ear fullness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
early satiety (Gastrointestinal disorders) | 2 (2) | 0 (0)
edema (Cardiac disorders) | 6 (6) | 4 (4)
elevated INR (Hepatobiliary disorders) | 19 (24) | 15 (16)
encephalopathy (Hepatobiliary disorders) | 11 (11) | 7 (7)
epistaxis (General disorders) | 3 (3) | 1 (1)
erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
face/mouth sensitivity (Nervous system disorders) | 1 (1) | 0 (0)
facial droop (Nervous system disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 22 (26) | 31 (37)
fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0)
fever (Infections and infestations) | 8 (10) | 2 (2)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
flu-like symptoms (General disorders) | 0 (0) | 1 (1)
gastritis (Infections and infestations) | 1 (2) | 2 (2)
gastrointestinal bleed (Gastrointestinal disorders) | 6 (6) | 3 (3)
gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
g.i disturbance (Gastrointestinal disorders) | 1 (1) | 0 (0)
glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1)
groin pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
gynecomastia (Hepatobiliary disorders) | 0 (0) | 2 (3)
hand-foot reaction (Skin and subcutaneous tissue disorders) | 25 (37) | 24 (36)
head cold (General disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 5 (5) | 7 (8)
hearing impairment (Ear and labyrinth disorders) | 0 (0) | 1 (1)
hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
hematuria with catherization (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
hemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (3)
hepatomegaly (Hepatobiliary disorders) | 2 (2) | 0 (0)
hiccups (Gastrointestinal disorders) | 2 (2) | 0 (0)
hypertension (Cardiac disorders) | 32 (56) | 29 (49)
hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
hyperkalemia (Renal and urinary disorders) | 4 (4) | 1 (1)
hypoalbuminemia (Hepatobiliary disorders) | 31 (43) | 27 (37)
hypokalemia (Renal and urinary disorders) | 6 (6) | 1 (1)
hypomagnesemia (Renal and urinary disorders) | 5 (8) | 5 (5)
hyponatremia (Renal and urinary disorders) | 1 (1) | 1 (1)
hypophosphatemia (Renal and urinary disorders) | 23 (37) | 23 (30)
hypotension (Cardiac disorders) | 2 (2) | 2 (2)
impaired speech (Nervous system disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 4 (4) | 6 (6)
irritability (Psychiatric disorders) | 1 (1) | 0 (0)
jaundice (Hepatobiliary disorders) | 1 (1) | 1 (1)
keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
left portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
liver failure (Hepatobiliary disorders) | 6 (6) | 5 (5)
leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
leukopenia (Blood and lymphatic system disorders) | 20 (29) | 11 (16)
lightheadedness (General disorders) | 2 (2) | 0 (0)
lipase elevation (Gastrointestinal disorders) | 22 (38) | 26 (49)
lymphodenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
mood alteration (Psychiatric disorders) | 1 (1) | 0 (0)
mucositis (Gastrointestinal disorders) | 0 (0) | 2 (2)
muscle cramps (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (11)
MRSA (Infections and infestations) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
nasal fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 21 (24) | 19 (20)
night sweats (General disorders) | 0 (0) | 1 (1)
nose tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
oral aphthous ulcers (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
oral hypersensitivity (Gastrointestinal disorders) | 1 (1) | 2 (2)
oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
oral thrush (Infections and infestations) | 0 (0) | 1 (1)
otitis media (Ear and labyrinth disorders) | 1 (1) | 0 (0)
palmer erythema (Hepatobiliary disorders) | 1 (1) | 0 (0)
palpitations (Cardiac disorders) | 0 (0) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
pelvic floor dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
perianal abcess (Gastrointestinal disorders) | 0 (0) | 1 (1)
peripheral neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
peritoneal enlarged studding (Gastrointestinal disorders) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 2 (2)
post-tace syndrome (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
poison ivy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
pseudogout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 12 (13) | 13 (18)
rectal fissue (Gastrointestinal disorders) | 0 (0) | 1 (1)
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
ringworm (Infections and infestations) | 1 (1) | 0 (0)
scalp hypersensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
sciatica (Nervous system disorders) | 1 (1) | 0 (0)
scortal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
seizure like activity (Nervous system disorders) | 1 (1) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
sinusitis (Infections and infestations) | 0 (0) | 2 (2)
skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
skin excoriation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
skin lesions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skull infection (Infections and infestations) | 0 (0) | 1 (1)
somnolence (Nervous system disorders) | 1 (1) | 1 (1)
spider angiomata (Hepatobiliary disorders) | 1 (1) | 0 (0)
spinal spondolytis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
splenomegaly (Hepatobiliary disorders) | 1 (1) | 2 (3)
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
stye (Infections and infestations) | 0 (0) | 1 (2)
systolic murmur (Cardiac disorders) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
temporal wasting (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
throat pain (Infections and infestations) | 2 (2) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 30 (41) | 26 (39)
thrush (Infections and infestations) | 1 (1) | 0 (0)
tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
tooth pain (General disorders) | 1 (1) | 0 (0)
total hyperbilirubinemia (Hepatobiliary disorders) | 32 (50) | 34 (53)
umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
unsteady gait (Nervous system disorders) | 3 (3) | 2 (2)
upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 2 (2) | 3 (4)
ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
vertigo (Nervous system disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 11 (11) | 9 (11)
weight loss (General disorders) | 40 (63) | 28 (39)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No